CLINICAL TRIAL: NCT02322983
Title: Effect Evaluation of Conscious Sedation With Nitrous Oxide at Control of Stress During Dental Care in Individuals With Cerebral Palsy.
Brief Title: Conscious Sedation With Nitrous Oxide in Control of Stress During Dental Care for Individuals With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cruzeiro do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fernando Martins Baeder, Researcher and professor of the degree program., Universidade Cruzeiro do Sul
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3307801700P7; CE/UCS - 044/2010 (Registry Identifier: Ethics and Research Committee of Unicsul)
Record Dates: First submitted 2014-12-13; First posted 2014-12-23 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Dental Care; Conscious Sedation; Autonomic Nervous System; Nitrous Oxide
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cerebral Palsy Subjects (Experimental): Use of conscious sedation with nitrous oxide in the control of stress during dental treatment in individuals with Cerebral Palsy
  Interventions: Behavioral: Control of Stress

INTERVENTIONS:
Behavioral: Control of Stress — To control stress were measured (at different times: T1, T2, T3 and T4) Venham's Score, Heart Rate, Respiratory Rate, and the titration of gases.

SUMMARY:
Cerebral Palsy induces oral alterations that impact on oral health, requiring dental treatment. The objective of this study was to evaluate the use of conscious sedation with nitrous oxide (N2O) in the control of stress during dental treatment in individuals with Cerebral Palsy.

DETAILED DESCRIPTION:
Were invited and accepted to participate in this study, 77 individuals with Cerebral Palsy who attended the outpatient clinic of San Francisco Home School (SFHS) at the time of data collection.

This study served as a non-randomized experimental trial conducted between 2011/2012 at dental ambulatory in the SFHS. Dental care routines have been established, by standardizing procedures and ensuring the reproducibility of the method of sedation. In the initial consultation, medical history taking (collecting sociodemographic data of the participants) and dental examination was performed. Data relating to the Cerebral Palsy clinical standard were collected from medical records of patients and noted in the evaluation sheet developed specifically for this research. Were provided to guardians the clarifications regarding sedation technique and treatment planning.

At dental examination the diagnostic criteria of caries followed those proposed by the World Health Organization (WHO). On the second visit, the patient was stabilized in the dental chair under mechanical contention. Performed adaptation and selection of nasal mask, monitoring equipment were positioned, starting the observation and recording of the behavioral and physiological records in the evaluation sheets. The proportion of gas was manipulated relative to the percentage between nitrous oxide and oxygen to achieve optimal sedation. In this study, it was considered a good sedation for Cerebral Palsy patient when he showed a certain degree of relaxation, which becomes more cooperative with treatment.

Behavioral assessment in relation to dental treatment was measured by Venham's Score, standard used for behavioral assessment of the dental patient, and the measurement performed according to the patient's behavior during the dental procedure.

Due to the subjectivity which compose the diagnosis of diseases or behavior analysis, it is common to occur some variation in the results. In the specific situation of a study, there is the aggravation of multiple observations be conducted on the same day, so that fatigue could lead to inconsistent diagnoses. For this reason, only one patient per day received dental care with nitrous oxide (N2O). In light of the above considerations, two dentists were calibrated to evaluate behavior in Venham's Score.

Behavioral and the physiological parameters evaluations of patients referred for dental treatment were performed in four stages: pre-sedation, induction, sedated patient and in the end.

Measures of Heart Rate and Respiratory Rate were recorded in all time intervals. The Heart Rate was later corrected for physiological cardiac variability in the different age groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy medical diagnosis;
* Age over 3 years old without distinction by gender;
* Patients with any clinical patterns of Cerebral Palsy;
* Patients with caries in at least two molars (primary or permanent), indicating anesthetic use for performing the restorative procedure.

Exclusion Criteria:

* Patients with chronic respiratory problems (such as chronic bronchitis, COPD) or acute (like flu with nasal congestion and active pneumonia) as these conditions contraindicate the use of N2O;
* Cerebral Palsy patients with genetic syndromes associated;
* Patients whose caregivers refused to sign the Instrument of Consent and the Consent of the Use of Conscious Sedation.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Heart Rate | data were collected and participants were followed up during dental care. An expected average of 1 hour.
Respiratory Rate | data were collected and participants were followed up during dental care. An expected average of 1 hour.
Venham's Score | data were collected and participants were followed up during dental care. An expected average of 1 hour.
Nitrous oxide and Oxygen Proportion | data were collected and participants were followed up during dental care. An expected average of 1 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando M Baeder, PhD, Principal Investigator — Universidade Cruzeiro do Sul
Locations (1):
- Universidade Cruzeiro do Sul, São Paulo, São Paulo, Brazil